CLINICAL TRIAL: NCT01620151
Title: A Randomized Controlled Trial Comparing Post-operative Pain & Outcomes of Open Thyroidectomy; Extended Neck vs No Extended Neck
Brief Title: Open Thyroid Surgery With Pillow Versus no Pillow for Better Post-operative Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Lang Hung Hin, Brian, Honorary Clinical Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RCTECS001
Record Dates: First submitted 2012-03-08; First posted 2012-06-15 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-12

CONDITIONS: Post-operative Pain
Keywords: Post-operative pain; Wound bleeding requiring exploration; PTH; RLN complication; Hypocalcaemia complication
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- No extended neck (No Intervention): Patient will not undergo thyroid surgery with extended neck
- Extended neck (Experimental): Patients who undergoing thyroid surgeries are positioned with extended neck by using pillow under shoulder in order to facilitate neck exposure and make the surgery easier.
  Interventions: Procedure: Extended neck with standard support or pillow

INTERVENTIONS:
Procedure: Extended neck with standard support or pillow — Patient will undergo thyroid surgery with an extended neck
  Other Names: neck extension; neck hyper-extension
  Arms: Extended neck

SUMMARY:
Primary: To compare the post-operative pain in patients with neck extension and without neck extension.

Secondary: To determine the benefit of neck exposure and peri-operative complications, which include duration of operation, intra-operative blood loss, recurrent nerve (RLN) injury and hypocalcaemia in both groups.

Hypothesis: Patients who undergoing thyroidectomy without neck extension will have less post-operative pain and there are no significant difference of post-operation complications between both groups.

DETAILED DESCRIPTION:
Conventional open thyroid surgery is still one of the most common operations performed globally. Traditionally, patients who undergoing thyroid surgeries are usually positioned with extended neck by using pillow under shoulder in order to facilitate neck exposure and make the surgery easier. However, the degree of benefit from the extended neck is doubtful and there is little objective evidence that suggest extended neck thyroid surgery offers better outcomes. On the the hand, over-extension of the neck should be avoided because of it is associated with post-operative pain, vomiting, spinal damage and stroke. The objective of the present study is to compare the post-operative pain in patients with neck extension and without neck extension. In addition to that, we also like to determine the benefit of neck exposure and peri-operative complications, which include duration of operation, intra-operative blood loss, recurrent nerve (RLN) injury and hypocalcaemia in both groups. This is a prospective randomized controlled trial, which will be conducted from 1st of March 2012 till 30th September 2012. Given that approximately 300 to 400 patients would undergo thyroid surgery in each year, we estimated 180 patients will be recruited and randomly divided into 2 groups (neck extension and no neck extension) before undergoing open thyroid surgery for this trial. Visual analogue scale (VAS) is used to determine the post-operative pain. Primary end point and other peri-operative variables are then analyzed with SPSS software.

ELIGIBILITY:
Inclusion Criteria:

* All patients who will be undergoing thyroid surgery in Queen Mary Hospital and Tung Wah Hospital.
* Age from 18 till 80 years old.

Exclusion Criteria:

* Patients with history of bleeding disorder and tendency.
* Patients with history of cervical spine surgery and disease.
* Patients with history of RLN injury and underlying cause of hypocalcemia.
* Patient with mental disorder and subnormal intelligence.
* Pregnant and lactating women.
* Patients who is having other surgical problem that needed other surgical procedure performed at the same setting.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2012-02; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Post-operative pain score | First postoperative week
  Post-operative pain ranges from 0 to 10 according to the Visual Analogue pain scale (VAS), and which 0 is 'No pain' and 10 is 'Worst possible pain'

SECONDARY OUTCOMES:
Surgically related complications | Immediate and after 6 months
  Neck exposure, duration of operation, skin incision length, intra-operative blood loss, RLN injury, post-operative hypocalcaemia
Postoperative pain scores | Day 0, day 1 and after two weeks
  Post-operative pain ranges from 0 to 10 according to the Visual Analogue pain scale (VAS), and which 0 is 'No pain' and 10 is 'Worst possible pain'

CONTACTS AND LOCATIONS:
Overall Officials: Hung Hin, Brian Lang, Dr., Principal Investigator — The University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong
  - Tung Wah Hospital, Sheung Wan

REFERENCES:
- [Background] Bae JS, Park WC, Song BJ, Jung SS, Kim JS. Endoscopic thyroidectomy and sentinel lymph node biopsy via an anterior chest approach for papillary thyroid cancer. Surg Today. 2009;39(2):178-81. doi: 10.1007/s00595-008-3840-5. Epub 2009 Feb 7. PMID 19199002
- [Background] Terris DJ, Bonnett A, Gourin CG, Chin E. Minimally invasive thyroidectomy using the Sofferman technique. Laryngoscope. 2005 Jun;115(6):1104-8. doi: 10.1097/01.MLG.0000163761.03764.44. PMID 15933531
- [Background] Park CS, Chung WY, Chang HS. Minimally invasive open thyroidectomy. Surg Today. 2001;31(8):665-9. doi: 10.1007/s005950170066. PMID 11510599
- [Background] Serpell JW, Grodski SF, O'Donell C. Does neck extension elevate the thyroid gland cephalad to potentially improve access during thyroidectomy? ANZ J Surg. 2003 Nov;73(11):887-9. doi: 10.1046/j.1445-2197.2003.02845.x. PMID 14616561
- [Background] Weintraub MI, Khoury A. Cerebral hemodynamic changes induced by simulated tracheal intubation: a possible role in perioperative stroke? Magnetic resonance angiography and flow analysis in 160 cases. Stroke. 1998 Aug;29(8):1644-9. doi: 10.1161/01.str.29.8.1644. PMID 9707207
- [Background] Lang BH, Lo CY. Total thyroidectomy for multinodular goiter in the elderly. Am J Surg. 2005 Sep;190(3):418-23. doi: 10.1016/j.amjsurg.2005.03.029. PMID 16105529
- [Background] Clements RH, Palepu R. In vivo comparison of the coagulation capability of SonoSurg and Harmonic Ace on 4 mm and 5 mm arteries. Surg Endosc. 2007 Dec;21(12):2203-6. doi: 10.1007/s00464-007-9345-2. Epub 2007 May 4. PMID 17479325
- [Background] Warden V, Hurley AC, Volicer L. Development and psychometric evaluation of the Pain Assessment in Advanced Dementia (PAINAD) scale. J Am Med Dir Assoc. 2003 Jan-Feb;4(1):9-15. doi: 10.1097/01.JAM.0000043422.31640.F7. PMID 12807591
- [Background] Beaver WT. Management of cancer pain with parenteral medication. JAMA. 1980 Dec 12;244(23):2653-7. No abstract available. PMID 7431615